CLINICAL TRIAL: NCT06195371
Title: The Impact of CASP3 Gene in Chemoresistant Breast Cancer
Brief Title: Impact of CASP3 Gene in Chemoresistance
Status: Not yet recruiting | Type: Observational
Sponsor: Gehad Salah El-Din shaker (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Gehad Salah El-Din shaker, Resident of clinical pathology department, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CASP3 gene in breast cancer
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. This study aims to evaluate the abnormalities of CASP3 gene in chemo resistance in breast cancer by FISH technique. evaluate the abnormalities of CASP3 gene in chemo resistance in breast cancer by FISH technique.
2. Detect CASP3 gene abnormality relation to survival, chemoresponse & chemoresistance.
3. Correlate CASP3 gene abnormalities with available clinicopathological data of breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common malignant tumor in women and the biggest threat to the health of women worldwide. Breast cancer represents a significant global health challenge: it is the most commonly diagnosed cancer in the world with an estimated 2.26 million cases recorded in 2020. Breast cancer is rarely seen in males. The incidence of breast cancer rises rapidly over the years, ranking as the first common cancer among females worldwide, and thus posing a considerable threat to female health. Breast cancer is the leading cause of cancer mortality among females. Although historically considered to be a disease of largely developed countries, over half of breast cancer diagnoses and two-thirds of breast cancer related deaths occurred in the less developed regions of the world in 2020.Being a highly prevalent cancer type, breast cancer is observed in both developing and developed countries with different causes and factors of progression. Adopting new life styles, industrialization, globalization, increased life expectancy, pollution etc are the leading causes of cancer. According to 2018 statistics, every year around 1.2 million new cases of breast cancer were diagnosed. The GLOBACON report of 2018 concluded that breast cancer was the most frequently identified cancer type and leading cause of cancer related death in majority of countries. Major part of breast related cancer is linked with the expression of estrogen receptors and their treatment is related with the disease prognosis. The rate of breast cancer mortality can be reduced down to a limit by early diagnosis; timely treatment and management . The commonly used chemotherapeutic drugs include doxorubicin (DOX), paclitaxel and cyclophosphamide. However, the efficiency of chemotherapy is greatly limited by primary and acquired drug resistance . Chemotherapy is widely accepted as traditional treatment method in spite of the obstacle of chemotherapy resistance. The important mechanisms that may lead to drug resistance include alteration in expression of ABC transporters gene family, damage of topoisomerase enzyme, mutation in DNA repair genes, induced apoptosis by genetic imbalance and alteration in signalling pathways of NF alpha etc. All these worsen the condition of breast cancer making chemotherapy a failure in most cases. According to Yaghoubi et al., 2015, the cells which already acquired drug resistance show cross resistance to anti proliferative nature of anti-oestrogen drugs which have crucial role in breast cancer treatment .Caspase-3, a cysteine-aspartic acid protease, has recently attracted much attention . Caspase-3 is a protein (also called CPP32 or apopain), encoded by the CASP3 gene; which is located in the 4q34 with size 2635 bp. It mediates apoptosis in response to chemotherapy, but losing caspase 3 activity causes cell survival and induces drug resistance through apoptotic pathway in breast cancer .Caspase-3 has been identified as a key mediator of apoptosis, activated in apoptotic cells by both extrinsic (death ligands) and intrinsic (mitochondrial) pathways. It also has several nonapoptotic functions such as involving in tissue differentiation, regeneration, and neural development. Nonconforming activation of caspase-3 can lead to tumorigenesis instead of inducing the programmed cell death.Recent progress in caspase research indicates that caspases-3 is a prominent enzyme not only in apoptotic flux but also in nonapoptotic processes such as tissue differentiation, tissue regeneration, and neural development.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients of breast cancer admitted to South Egypt Cancer Institute at different stages of the disease

Exclusion Criteria:

* Other malignant diseases-Male breast cancer .

Ages: 15 Years to 75 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: female patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
- Evaluation of casp3 gene abnormalities by fluorescence in situ hybridization in patients with breast cancer | baseline
  Evaluation of casp3 gene abnormalities by fluorescence in situ hybridization in patients with breast cancer

SECONDARY OUTCOMES:
- correlation between casp3 gene and response to Chemotherapy. | baseline
  correlation between casp3 gene and response to Chemotherapy.

REFERENCES:
- [Background] Fu W, Song J, Li H. Breviscapine reverses doxorubicin resistance in breast cancer and its related mechanisms. Thorac Cancer. 2023 Sep;14(27):2785-2792. doi: 10.1111/1759-7714.15072. Epub 2023 Aug 16. PMID 37584258
- [Background] Wilkinson L, Gathani T. Understanding breast cancer as a global health concern. Br J Radiol. 2022 Feb 1;95(1130):20211033. doi: 10.1259/bjr.20211033. Epub 2021 Dec 14. PMID 34905391
- [Background] Xu F, Xia T, Xu QT, Zhang X, Huang YZ, Sun X, Shi L, Zhou XJ, Wei JF, Ding Q. RBMS2 Chemosensitizes Breast Cancer Cells to Doxorubicin by Regulating BMF Expression. Int J Biol Sci. 2022 Feb 7;18(4):1724-1736. doi: 10.7150/ijbs.66480. eCollection 2022. PMID 35280673
- [Background] Yaghoubi A, Ghojazadeh M, Abolhasani S, Alikhah H, Khaki-Khatibi F. Correlation of Serum Levels of Vitronectin, Malondialdehyde and Hs- CRP With Disease Severity in Coronary Artery Disease. J Cardiovasc Thorac Res. 2015;7(3):113-7. doi: 10.15171/jcvtr.2015.24. PMID 26430499
- [Background] Asadi M, Taghizadeh S, Kaviani E, Vakili O, Taheri-Anganeh M, Tahamtan M, Savardashtaki A. Caspase-3: Structure, function, and biotechnological aspects. Biotechnol Appl Biochem. 2022 Aug;69(4):1633-1645. doi: 10.1002/bab.2233. Epub 2021 Aug 22. PMID 34342377
- [Background] Jakubowska K, Guzinska-Ustymowicz K, Famulski W, Cepowicz D, Jagodzinska D, Pryczynicz A. Reduced expression of caspase-8 and cleaved caspase-3 in pancreatic ductal adenocarcinoma cells. Oncol Lett. 2016 Mar;11(3):1879-1884. doi: 10.3892/ol.2016.4125. Epub 2016 Jan 19. PMID 26998093
- [Background] Shalini S, Dorstyn L, Dawar S, Kumar S. Old, new and emerging functions of caspases. Cell Death Differ. 2015 Apr;22(4):526-39. doi: 10.1038/cdd.2014.216. Epub 2014 Dec 19. PMID 25526085